CLINICAL TRIAL: NCT06533670
Title: Tumor Microenvironment Alteration During Neoadjuvant Chemotherapy in HER2 Positive Breast Cancer Patients
Brief Title: TME Alteration in HER2 Positive Breast Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Wonshik Han, Professor, Seoul National University Hospital
Other Study IDs: 2402-110-1514
Record Dates: First submitted 2024-07-30; First posted 2024-08-01 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; HER2-positive Breast Cancer; Chemotherapy Effect
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluate for changes in the tumor microenvironment before/during neoadjuvant chemotherapy and after treatment in patients diagnosed with HER2-positive advanced breast cancer and receiving neoadjuvant cancer therapy and surgery for curative purposes.

ELIGIBILITY:
Inclusion criteria i. Adult patients over 18 years of age ii. Patients undergoing curative treatment including neoadjuvant chemotherapy after confirmation of breast cancer without distant metastases iii. Clinical T stage II-IV patients iv. HER2 positive breast cancer patients

Exclusion criteria If you have other comorbidities that, according to the researcher's judgment, may affect the results of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HER2 positive breast cancer patients undergoing curative treatment including neoadjuvant chemotherapy after confirmation of breast cancer without distant metastases
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-07-19 (Actual); Primary Completion 2026-07-19 (Estimated); Study Completion 2026-07-19 (Estimated)

PRIMARY OUTCOMES:
tumor microenvironment alteration | 6 months
  tumor microenvironment changes during neoadjuvant chemotherapy (NAC) for HER2-positive breast cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea